CLINICAL TRIAL: NCT07396207
Title: The Effect of a Gamified Metaverse-Based Education on Nursing Students' Knowledge and Attitudes Toward Ventrogluteal Intramuscular Injection
Brief Title: Gamified Metaverse Education for Ventrogluteal IM Injection (G-META-IM)
Acronym: G-META-IM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Aliye Yıldırım, Investigator, Baskent University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: E-62310886-605-543580
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Nursing Education; Intramuscular Injection; Metaverse
Keywords: Metaverse; Intramuscular Injection; Nursing education

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to either an intervention group receiving a gamified, metaverse-based education program or a control group receiving traditional education, and outcomes will be compared between the two parallel groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metaverse-Based Gamified Education (Experimental): Participants in this arm will receive a gamified, metaverse-based education program designed to teach ventrogluteal intramuscular injection, including anatomical landmark identification using the V method and correct injection procedures.
  Interventions: Behavioral: Gamified Metaverse-Based Education Program
- Traditional Education (No Intervention): Participants in this arm will receive traditional education on ventrogluteal intramuscular injection delivered using standard teaching methods commonly used in nursing education.

INTERVENTIONS:
Behavioral: Gamified Metaverse-Based Education Program — Standard theoretical instruction on ventrogluteal intramuscular injection delivered using conventional teaching methods commonly used in nursing education.
  Other Names: Metaverse-Based Gamified Education
  Arms: Metaverse-Based Gamified Education

SUMMARY:
This study aims to examine the effect of a gamified, metaverse-based education program on nursing students' knowledge and attitudes regarding ventrogluteal intramuscular injection. Intramuscular injection is a commonly used nursing skill that requires accurate anatomical knowledge and correct technique to ensure patient safety. The ventrogluteal site is considered a safe injection site; however, nursing students often report limited knowledge and confidence in its use.

In this study, nursing students will be assigned to either an intervention group or a control group. The intervention group will receive a gamified metaverse-based educational program designed to teach ventrogluteal site identification using the V method and the correct steps of intramuscular injection. The control group will receive traditional education using standard teaching methods.

Data will be collected before and after the educational intervention using a knowledge test and a learning attitude scale. The results of this study are expected to provide evidence on the effectiveness of metaverse-based and gamified education approaches in nursing education and to support the development of safe and innovative learning environments for nursing students.

DETAILED DESCRIPTION:
This study is designed to evaluate the effectiveness of a gamified, metaverse-based educational program on nursing students' knowledge and attitudes toward ventrogluteal intramuscular (IM) injection. Intramuscular injection is a fundamental nursing skill that requires accurate identification of anatomical landmarks and adherence to safe injection principles. Although the ventrogluteal site is recommended as a safe injection site due to its anatomical advantages, its use remains limited among nursing students, often due to insufficient knowledge, lack of confidence, and limited practical experience.

The study will be conducted using a quasi-experimental design with an intervention group and a control group. The study population will consist of first-year nursing students enrolled in a nursing program during the 2025-2026 academic year. Eligible participants who provide informed consent will be assigned to either the intervention group or the control group.

The intervention group will receive a gamified metaverse-based education program developed to support learning of ventrogluteal site anatomy, identification of the injection site using the V method, and the correct steps of intramuscular injection. The program includes interactive virtual learning modules, educational videos, and game-based assessment activities designed to enhance engagement and learning motivation. The control group will receive traditional education delivered through standard teaching methods commonly used in nursing education.

Data will be collected from both groups before and after the educational intervention. Data collection tools will include a sociodemographic information form, a knowledge test related to ventrogluteal intramuscular injection, and a learning attitude scale. Pre-intervention and post-intervention measurements will be compared to assess changes in knowledge levels and learning attitudes between and within groups.

The findings of this study are expected to contribute to the growing body of evidence on the use of digital, immersive, and gamified learning approaches in nursing education. The results may support the integration of metaverse-based educational strategies into nursing curricula and help improve safe injection practices by enhancing students' knowledge, confidence, and attitudes toward learning.

ELIGIBILITY:
Inclusion Criteria:

* Being enrolled as a first-year nursing student during the 2025-2026 academic year
* Having no prior formal education or training specifically focused on ventrogluteal intramuscular injection
* Willingness to participate in the study
* Providing written informed consent

Exclusion Criteria:

* Previous participation in a structured training or simulation program related to ventrogluteal intramuscular injection
* Incomplete participation in the educational intervention or data collection process
* Declining or withdrawing informed consent at any stage of the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Knowledge Level Regarding Ventrogluteal Intramuscular Injection | Before and immediately after the educational intervention
  The level of knowledge of nursing students regarding ventrogluteal intramuscular injection, including anatomical landmark identification and correct injection procedures, measured using a structured knowledge test.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cetinkaya Uslusoy E, Aydinli A, Durna F. Enhancing learning motivation and academic achievement in nursing students through metaverse-based learning: A randomized controlled study. Jpn J Nurs Sci. 2024 Jul;21(3):e12594. doi: 10.1111/jjns.12594. Epub 2024 Feb 29. PMID 38425133